CLINICAL TRIAL: NCT00270023
Title: Recombinant Human Erythropoietin (R-HuEPO) in Non-Anemic Patients Scheduled for Selective Orthopedic and Vascular Surgery or Reductive Mammoplasty to Facilitate Presurgical Autologous Blood Donation Combined With Normo-Volemic Hemodilution (NVHD)
Brief Title: A Study to Determine the Effectiveness of Epoetin Alfa in Facilitating Self-donation of Blood Before Surgery in Non-anemic Patients Who Are Undergoing Orthopedic, Heart and Blood Vessel, or Breast Reduction Surgery; Performed in Combination With a Procedure to Reduce Blood Loss During Surgery.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR005890
Record Dates: First submitted 2005-12-22; First posted 2005-12-26 (Estimated); Last update posted 2011-05-18 (Estimated); Status verified 2010-04

CONDITIONS: Blood Transfusion; Blood Transfusion, Autologous; Orthopedic Procedures; Orthopedic Surgery; Cardiovascular Surgical Procedures; Mammaplasty
Keywords: Blood transfusion; epoetin alfa; epogen; erythropoietin; orthopedic procedures; orthopedic surgery; cardiovascular surgical procedures; breast reduction
MeSH Terms: interventions — Epoetin Alfa

INTERVENTIONS:
Drug: epoetin alfa

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of epoetin alfa and whether epoetin alfa will enable self-donation of blood during an 11-day period before surgery (which is shorter than the conventional 3-week blood donation period before surgery) in patients who are not anemic and who will be undergoing orthopedic, heart and blood vessel, or breast reduction surgery. Epoetin alfa is a genetically engineered protein that stimulates red blood cell production. Normovolemic hemodilution (NVHD, withdrawal of a patient's blood immediately before surgery, immediate replacement of blood with an equal volume of fluid, and return of the withdrawn blood after completion of surgery; a procedure which reduces the loss of blood during surgery) will also be performed.

DETAILED DESCRIPTION:
Patients undergoing surgery frequently require blood transfusions both during and after the operation. Patients often have their own blood collected for this purpose over a standard 3- to 4-week presurgical period. However, a large percentage of patients are not able to pre-donate their own blood for transfusion. Agents that can facilitate self-donation in less time than the conventional 3 weeks before surgery and reduce the need for transfusions from others, may improve the overall safety of surgery. This is a randomized, double-blind, placebo-controlled, parallel group, multicenter study to determine whether epoetin alfa will enable the self-donation of at least 4 units of blood in the shortened presurgical time period of 11 days before surgery (which is a shorter period of time than the conventional 3 week blood donation period before surgery) in patients who are not anemic and who are undergoing orthopedic, heart and blood vessel, or breast reduction surgery. The study consists of a 7-day screening period during which patients will be tested for eligibility for the study; an 11-day treatment, blood collection, and evaluation period that ends on Day 11 (the day of surgery); and a post-surgery follow-up period beginning on the evening of Day 11 and ending with a final study visit at the time a patient is discharged from the hospital after surgery. Patients will be randomly assigned to one of four treatment groups: epoetin alfa 300 units/kilogram (U/kg), epoetin alfa 600 U/kg, placebo to match the volume of epoetin alfa 300 U/kg, or placebo to match the volume of epoetin alfa 600 U/kg, given by injection into a vein. Twice as many patients will receive treatment with epoetin alfa as will receive treatment with placebo. A total of 3 doses of study drug will be administered before surgery; one dose will be given on each of Days 1, 4, and 7 of the study. Additionally, from Day 1 to the day of hospital discharge, all patients will receive 200 milligrams of iron and 5 milligrams of a folate supplement daily by mouth to help the body to increase the production of red blood cells. On Day 1, before the first dose of study medication, one unit of blood will be collected from each patient and stored for self-donated blood transfusion. An additional unit of blood will be obtained from each patient (before the administration of study drug) and stored for self-donated blood transfusion on each of Days 4, 7, and 11 (the day of surgery, before the operation); this will only be performed if the patient's hemoglobin is >11.0 g/dL. If a patient's hemoglobin is lower than 11.0 g/dL, no blood will be collected from that patient on these days, although study drug will continue to be given. Normovolemic hemodilution (NVHD) will be performed on Day 11, the day of surgery, before and during the operation. Safety evaluations include laboratory tests, vital signs, and the recording of adverse events. Effectiveness will be assessed by comparing the number of self-donated units of blood obtained within 11 days among the 4 treatment groups, and secondarily by comparing the change in hemoglobin, immature red blood cells, and erythropoietin (the red blood cell stimulating hormone) levels in the blood among the 4 treatment groups from before the start of study to the end of the study. The study hypothesis is that in an abbreviated time period before surgery (11 days), epoetin alfa will stimulate the generation of 4 units of self-donated blood in patients who are not anemic who are undergoing orthopedic, heart and blood vessel, or breast reduction surgery. Epoetin alfa 300 units/kilogram (U/kg), epoetin alfa 600 U/kg, or placebo, by injection into a vein; given on each of Days 1, 4, and 7 of the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients scheduled for orthopedic surgery, heart and blood vessel surgery, or breast reduction surgery
* having an anticipated requirement of 3 or more units of blood
* who are non-anemic (hemoglobin within normal range of 12.0 - 18.0 grams/deciliter)
* having laboratory tests within normal ranges

Exclusion Criteria:

* Patients with history of any blood disease
* having signs and symptoms of significant disease/dysfunction
* having uncontrolled high blood pressure or signs and symptoms of significant dizziness, faintness, or lightheadedness which appear only on standing, and which are caused by low blood pressure
* who have received a blood transfusion within 1 month before the start of the study
* having a body weight >100 kilograms (approximately 220 pounds)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Study Completion 1991-11 (Actual)

PRIMARY OUTCOMES:
Number of self-donated units of blood obtained within 11 days; Assessment of safety (laboratory tests, vital signs, and adverse events) from before the study to the end of the study

SECONDARY OUTCOMES:
Changes in hemoglobin, reticulocytes (immature red blood cells), and erythropoietin (red blood cell stimulating hormone) levels in blood from before the study to the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study to determine the effectiveness of epoetin alfa in facilitating self-donation of blood before surgery in non-anemic patients scheduled for selective orthopedic, vasucular, or breast reduction surgery — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=676&filename=CR005890_CSR.pdf